CLINICAL TRIAL: NCT07091266
Title: A Prospective Randomized Controlled Trial Comparing the Therapeutic Efficacy of Sacral Neuromodulation Versus Hyperbaric Oxygen Therapy in Patients With Refractory Interstitial Cystitis and Bladder Pain Syndrome
Brief Title: SNM vs. HBOT for Refractory IC/BPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyan City Renmin Hospital (Other Government)
Responsible Party: Principal Investigator, Yan Wen, Principal investigator, Shiyan City Renmin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2020-K056
Record Dates: First submitted 2025-07-11; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Interstitial Cystitis/Bladder Pain Syndrome; Underactive Bladder
MeSH Terms: conditions — Cystitis, Interstitial; Urinary Bladder, Underactive | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Sacral Neuromodulation (SNM) Group (Experimental): Patients were randomized to receive sacral neuromodulation therapy. They were followed up at 1 month and 3 months post-procedure.
  Interventions: Device: Sacral Neuromodulation (SNM)
- Active Comparator: Hyperbaric Oxygen Therapy (HBOT) Group (Active Comparator): Patients were randomized to receive hyperbaric oxygen therapy. They were followed up at 1 month and 3 months post-treatment.
  Interventions: Procedure: Hyperbaric Oxygen Therapy (HBOT)

INTERVENTIONS:
Device: Sacral Neuromodulation (SNM) — A standardized two-stage implantation protocol was used. In Stage 1, a temporary lead (InterStim 3093, Medtronic) was implanted at the S3 sacral foramen under fluoroscopic guidance. Patients with ≥50% improvement in urinary symptoms over a 7-day test period proceeded to Stage 2, where a permanent neurostimulator (InterStim 3058, Medtronic) was implanted subcutaneously. Stimulation parameters were adjusted (amplitude: 0.5-10 V; frequency: 14 Hz; pulse width: 210 μs) to optimize symptom control.
  Arms: Experimental: Sacral Neuromodulation (SNM) Group
Procedure: Hyperbaric Oxygen Therapy (HBOT) — Patients received two 20-session courses (5 sessions/week) in a hyperbaric chamber at 2.0 atmospheres absolute (ATA). Each session consisted of 60 minutes of 100% oxygen inhalation, bracketed by compression and decompression periods.
  Arms: Active Comparator: Hyperbaric Oxygen Therapy (HBOT) Group

SUMMARY:
This study is for people with long-term bladder pain and urinary problems (known as Interstitial Cystitis/Bladder Pain Syndrome or IC/BPS) that have not improved with other treatments. The study compares two different treatments: Sacral Neuromodulation (SNM), which uses an implanted device to send gentle electrical pulses to nerves controlling the bladder, and Hyperbaric Oxygen Therapy (HBOT), where patients breathe pure oxygen in a special chamber. Participants were randomly assigned to one of the two groups to help doctors understand which treatment works better to reduce symptoms and improve quality of life.

DETAILED DESCRIPTION:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a chronic, debilitating condition that is often refractory to conventional treatments. Sacral neuromodulation (SNM) is a third-line therapy recognized by AUA/EAU guidelines, while hyperbaric oxygen therapy (HBOT) is an emerging treatment with potential anti-inflammatory benefits. There is a lack of direct comparative evidence between these two modalities. This study prospectively enrolled and randomized 88 patients with refractory IC/BPS to receive either SNM (study group) or HBOT (control group). The primary objective is to compare changes in urinary symptoms, urodynamic parameters, and quality of life scores between the two groups at baseline, 1-month, and 3-month follow-ups. The study aims to provide robust evidence to guide treatment selection for refractory IC/BPS patients who have failed at least two prior therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosis of refractory Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) according to AUA/SUFU guidelines, confirmed by cystoscopy with hydrodistention and glomerulations, and/or Hunner's lesions.
* Failure of at least two prior therapies (e.g., oral medications, intravesical instillations, pelvic floor physical therapy).
* Willingness to provide written informed consent.

Exclusion Criteria:

* Presence of urinary tract malignancies, pelvic organ prolapse ≥ stage III, or urethral stricture.
* Low-compliance bladder (<10 mL/cm H₂O), organic bladder outlet obstruction, or active urinary tract infection.
* Contraindications to surgery (e.g., coagulopathy, existing pacemaker) or HBOT (e.g., untreated pneumothorax).
* Pregnancy.
* Presence of psychiatric disorders or inability to comply with follow-up protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Daily Urination Frequency | Baseline, 1 Month, 3 Months
  Measured by a 3-day bladder diary as the average number of voids per 24 hours. A lower value indicates better outcome.
Change in Nocturia Frequency | Baseline, 1 Month, 3 Months
  Measured by a 3-day bladder diary as the average number of nighttime voids. A lower value indicates better outcome.
Change from Baseline in Quality of Life Score at 3 Months | Baseline, 3 Months
  Measured using the Incontinence Quality of Life Questionnaire-Short Form (ICI-Q-SF). A lower score indicates better quality of life.
Change in Pain Severity | Baseline, 1 Month, 3 Months
  Measured using a Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Change in Post-void Residual (PVR) Volume | Baseline, 1 Month, 3 Months
  Measured by ultrasound in milliliters (mL).
Change in Maximum Voided Volume (MVV) | Baseline, 1 Month, 3 Months
  Measured by a 3-day bladder diary in milliliters (mL).
Change in Average Voided Volume (AVV) | Baseline, 1 Month, 3 Months
  Measured by a 3-day bladder diary in milliliters (mL).
Change in Bladder Compliance (BC) | Baseline, 1 Month, 3 Months
  Measured via urodynamic studies as the change in bladder volume per unit change in pressure. Unit: milliliters per centimeter of water (mL/cm H₂O).
Change in Maximum Urethral Closure Pressure (MUCP) | Baseline, 1 Month, 3 Months
  Measured via urodynamic studies to assess urethral sphincter function. Unit: centimeters of water (cm H₂O).
Change in Abdominal Leak Point Pressure (ALPP) | Baseline, 1 Month, 3 Months
  Measured via urodynamic studies as the intravesical pressure at which urine leakage occurs during a cough or strain. Unit: centimeters of water (cm H₂O).
Incidence of Adverse Events | Up to 3 months
  Number of participants experiencing adverse events, such as pain at the implantation site, symptom recurrence, electrode displacement, urinary tract infection, dizziness, or vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital, Hubei University of Medicine, Shiyan, Hubei, China